CLINICAL TRIAL: NCT01106859
Title: Assessment of Next-Morning Driving Performance After Middle of the Night Administration of Zolpidem Tartrate Sublingual Tablet 3.5 mg in Healthy Adult Volunteers: Single-center, Double-blind, Randomized, Placebo-controlled, Four-way Crossover Study
Brief Title: Driving Performance After Middle of the Night Administration of 3.5 mg Zolpidem Tartrate Sublingual Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Transcept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ZI-18; 2010-019959-22 (EudraCT Number)
Record Dates: First submitted 2010-04-16; First posted 2010-04-20 (Estimated); Results first posted 2012-01-20 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Insomnia
Keywords: insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — zopiclone; Zolpidem; Administration, Sublingual

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- zopiclone (Active Comparator): Zopiclone is taken at bedtime 9 hours before driving. The middle-of-the-night medication is a placebo matching zolpidem tartrate sublingual tablet.
  Interventions: Drug: zopiclone; Drug: Placebo (sublingual tablet)
- zolpidem 3 hours prior (Experimental): A placebo matching zopiclone is taken at bedtime. The middle-of-the-night treatment is zolpidem tartrate sublingual tablet taken 3 hours prior to driving.
  Interventions: Drug: zolpidem tartrate sublingual tablet; Drug: Placebo
- zolpidem 4 hours prior (Experimental): A placebo matching zopiclone is taken at bedtime. The middle-of-the-night treatment is zolpidem tartrate sublingual tablet taken 4 hours prior to driving.
  Interventions: Drug: zolpidem tartrate sublingual tablet; Drug: Placebo
- Placebo (Placebo Comparator): A placebo matching zopiclone is taken at bedtime. The middle-of-the-night treatment is a placebo matching zolpidem tartrate sublingual tablet.
  Interventions: Drug: Placebo (sublingual tablet); Drug: Placebo

INTERVENTIONS:
Drug: zopiclone — 7.5 mg tablet by mouth. Zopiclone is a commonly used hypnotic in Europe that is known to impair driving in the morning 9 hours after dosing.
  Other Names: non-benzodiazepine hypnotic agent; Zimovane; Imovane
  Arms: zopiclone
Drug: zolpidem tartrate sublingual tablet — 3.5 mg zolpidem tartrate sublingual tablet taken either 3 or 4 hours prior to driving. Participants placed the study drug under the tongue and allowed it to dissolve there for about 2 minutes, then swallowed after dissolved.
  Other Names: Intermezzo®
  Arms: zolpidem 3 hours prior; zolpidem 4 hours prior
Drug: Placebo (sublingual tablet) — Placebo matching zolpidem tartrate sublingual tablet taken either 3 or 4 hours prior to driving. Participants placed the study drug under the tongue and allowed it to dissolve there for about 2 minutes, then swallowed after dissolved.
  Arms: Placebo; zopiclone
Drug: Placebo — Placebo matching zopiclone
  Arms: Placebo; zolpidem 3 hours prior; zolpidem 4 hours prior

SUMMARY:
A study in healthy volunteers of the next morning driving performance after middle-of-the-night dosing of 3.5 mg zolpidem tartrate sublingual tablet, a sleep aid. The next morning driving performance will be measured by taking a standardized driving test.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 21 and 64 inclusive. For female subjects only: Female subjects will be included if they are post-menopausal or sterilized, or if they are of childbearing potential, they are not breastfeeding, their pregnancy test is negative, they have no intention of becoming pregnant during the course of the study, and are using adequate contraceptive drugs or devices. Medically acceptable methods of contraception that may be used by the subject and/or her partner are: oral contraceptives, progestin injection or implants, condom with spermicide, diaphragm with spermicide, IUD, vaginal spermicidal suppository, surgical sterilization or abstinence. Females using oral contraception must have started using the medication at least 4 weeks prior to screening. Surgical sterilization must have occurred at least 6 weeks prior to screening.
* Good health on the basis of pre-study history and physical examination, vital signs and the results of blood chemistry, hematology, and urinalysis
* Good binocular visual acuity, corrected or uncorrected
* Possession of valid driver's license for 3 years or more
* Driving experience at least 3000 km/year
* Signed informed consent

Exclusion Criteria:

* A history of drug addiction or drug or substance abuse, including alcohol abuse, within the past 12 months
* Has a history of restless legs syndrome, sleep apnea, narcolepsy or other primary sleep disorder
* A known hypersensitivity to zolpidem or zopiclone
* Has undergone oral surgery, tooth extraction or piercing of the lip/tongue within 60 days prior to screening
* Has used any medication to promote sleep, including herbal medications, within 14 days (or 5 half-lives of the drug, whichever is longer) prior to screening
* Prescription medications for other health conditions are allowed as long as the subject has been on a stable dose at least 30 days prior to screening
* Has taken any drugs known to induce hepatic drug metabolism (i.e., rifampin) within 30 days prior to screening
* BMI > 29 Kg/M^2
* Current use of medication that affects driving performance
* Smokes more than 10 cigarettes/day
* Uses tobacco products during periods of nighttime awakening
* Consumes more than 6 cups of coffee/day
* Consumes more than 21 glasses of alcohol/week
* Has received an investigational drug within 60 days or 5 half-lives (whichever is longer) prior to screening
* Has any additional condition(s) that in the Investigator's opinion would:

  * Affect sleep/wake function
  * Prohibit the subject from completing the study
  * Not be in the best interest of the subject to participate in the study

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annemiek Vermeeren, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] Vermeeren A, Vuurman EF, Leufkens TR, Van Leeuwen CJ, Van Oers AC, Laska E, Rico S, Steinberg F, Roth T. Residual effects of low-dose sublingual zolpidem on highway driving performance the morning after middle-of-the-night use. Sleep. 2014 Mar 1;37(3):489-96. doi: 10.5665/sleep.3482. PMID 24587571

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-four candidates were screened. Four screening failures: high blood pressure (2), positive drug test (1), personal reasons (1)
Groups:
- Total Population: All participants in this four-way cross-over study
Period: Overall Study
Arm/Group | Total Population
Started | 40 (Intent to treat population and safety population are the same (40 participants))
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Population
Number analyzed (Participants) | 40
Age Continuous [Mean (Standard Deviation); unit: years] | 37 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 39
  Black | 0
  Asian | 0
  Other | 1
Region of Enrollment [Number; unit: participants]
  Netherlands | 40
Height [Mean (Standard Deviation); unit: centimeters] | 176 (9)
Weight [Mean (Standard Deviation); unit: kilograms]
  Male | 79 (8)
  Female | 65 (8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/meter^2] | 23.2 (2.4)

OUTCOME MEASURES:

1. Secondary Outcome: Mean Standard Deviation of Lateral Position (SDLP) in the Highway Driving Test
Description: Standard deviation of lateral position (SDLP) in a highway-driving lane is a surrogate measure for driving performance. It measures the driver's ability to stay in a constant position within the driving lane. Variations in the lateral position are recorded and analyzed.
Time Frame: 3-9 hours post dose
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: centimeters
Groups:
- Zolpidem 4 Hours Prior: A placebo matching zopiclone is taken at bedtime. The middle-of-the-night treatment is 3.5 mg zolpidem tartrate sublingual tablet taken 4 hours prior to driving.
- Zolpidem 3 Hours Prior: A placebo matching zopiclone is taken at bedtime. The middle-of-the-night treatment is 3.5 mg zolpidem tartrate sublingual tablet taken 3 hours prior to driving.
- Zopiclone: Zopiclone (7.5 mg tablet) is taken at bedtime 9 hours before driving. The middle-of-the-night medication is a placebo matching zolpidem tartrate sublingual tablet.
Arm/Group | Zolpidem 4 Hours Prior | Zolpidem 3 Hours Prior | Zopiclone | Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40
centimeters | 16.7 (0.60) | 17.3 (0.60) | 18.3 (0.60) | 15.9 (0.60)
Statistical Analysis 1: Comparison: Zolpidem 4 Hours Prior vs Placebo; P-value is based on ANOVA model with fixed effects for sequence, period and treatment, a random effect for subject within sequence, and assuming compound symmetry covariance structure; the p-value is reported from LS Mean difference between Treatment Groups: LS mean of SDLP (Zolpidem 4 Hours) - LS mean of SDLP (Placebo); Test type: Superiority or Other; p = 0.0174, ANOVA — No p-value adjustment for multiple comparisons; The degrees of freedom are 114 for the p-value testing the difference between treatment groups; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [0.1 to 1.5]
Statistical Analysis 2: Comparison: Zolpidem 3 Hours Prior vs Placebo; P-value is based on ANOVA model with fixed effects for sequence, period and treatment, a random effect for subject within sequence, and assuming compound symmetry covariance structure; the p-value is reported from LS Mean difference between Treatment Groups: LS mean of SDLP (Zolpidem 3 Hours) - LS mean of SDLP (Placebo); Test type: Superiority or Other; p < 0.0001, ANOVA — No p-value adjustment for multiple comparisons; The degrees of freedom are 114 for the p-value testing the difference between treatment groups; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [0.8 to 2.1]
Statistical Analysis 3: Comparison: Zopiclone vs Placebo; P-value is based on ANOVA model with fixed effects for sequence, period and treatment, a random effect for subject within sequence, and assuming compound symmetry covariance structure; the p-value is reported from LS Mean difference between Treatment Groups: LS mean of SDLP (Zopiclone) - LS mean of SDLP (Placebo); Test type: Superiority or Other; p < 0.0001, ANOVA — No p-value adjustment for multiple comparisons; The degrees of freedom are 114 for the p-value testing the difference between treatment groups; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [1.8 to 3.1]

2. Secondary Outcome: Mean Standard Deviation of Speed (SDS) in the Highway Drive Test
Description: Mean standard deviation of speed (SDS) is a common measure of the driver's ability to maintain a constant driving speed. Variations in driving speed are recorded and analyzed.
Time Frame: 3-9 hours post dose
Population: Intent to treat population. In one Zopiclone case, the velocity of the car was not recorded due to technical problems, and therefore SDS could not be calculated in this drive.
Measure: Least Squares Mean (Standard Error); unit: kilometers/hour
Arm/Group | Zolpidem 4 Hours Prior | Zolpidem 3 Hours Prior | Zopiclone | Placebo
Number analyzed (Participants) | 40 | 40 | 39 | 40
kilometers/hour | 1.98 (0.08) | 1.91 (0.08) | 1.99 (0.08) | 1.83 (0.08)
Statistical Analysis 1: Comparison: Zolpidem 4 Hours Prior vs Placebo; P-value is based on ANOVA model with fixed effects for sequence, period and treatment, a random effect for subject within sequence, and assuming compound symmetry covariance structure; the p-value is reported from LS Mean difference between Treatment Groups: LS mean of SDS (Zolpidem 4 hours prior) - LS mean of SDS (Placebo); Test type: Superiority or Other; p = 0.0145, ANOVA — No p-value adjustment for multiple comparisons; The degrees of freedom are 113 for the p-value testing the difference between treatment groups; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.03 to 0.27]
Statistical Analysis 2: Comparison: Zolpidem 3 Hours Prior vs Placebo; P-value is based on ANOVA model with fixed effects for sequence, period and treatment, a random effect for subject within sequence, and assuming compound symmetry covariance structure; the p-value is reported from LS Mean difference between Treatment Groups: LS mean of SDS (Zolpidem 3 Hours) - LS mean of SDS (Placebo); Test type: Superiority or Other; p = 0.2179, ANOVA — No p-value adjustment for multiple comparisons; The degrees of freedom are 113 for the p-value testing the difference between treatment groups; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.05 to 0.20]
Statistical Analysis 3: Comparison: Zopiclone vs Placebo; P-value is based on ANOVA model with fixed effects for sequence, period and treatment, a random effect for subject within sequence, and assuming compound symmetry covariance structure; the p-value is reported from LS Mean difference between Treatment Groups: LS mean of SDS (Zopiclone) - LS mean of SDS (Placebo); Test type: Superiority or Other; p = 0.0096, ANOVA — No p-value adjustment for multiple comparisons; The degrees of freedom are 113 for the p-value testing the difference between treatment groups; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [0.04 to 0.29]

3. Secondary Outcome: Summary of Participants With Treatment Emergent Adverse Experiences (TEAEs)
Description: Adverse Events were graded by the investigator using the World Health Organization (WHO) Adverse Event Grading Scale and were assessed for severity (mild, moderate, severe) and relatedness (summarized as 'unrelated' and 'related') to study treatment. Also included are counts of participants with serious AEs, AEs leading to discontinuation of study treatment, and deaths.
Time Frame: Day 1 -6 weeks
Population: Safety population (participants who were randomized and received at least one dose of study drug)
Measure: Number; unit: participants
Arm/Group | Zolpidem 4 Hours Prior | Zolpidem 3 Hours Prior | Zopiclone | Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40
participants
  At least one TEAE | 5 | 5 | 6 | 4
  TEAE graded as mild | 4 | 5 | 6 | 4
  TEAE graded as moderate | 1 | 0 | 0 | 0
  TEAE graded as severe | 0 | 0 | 0 | 0
  Unrelated | 3 | 2 | 4 | 1
  Related | 2 | 3 | 2 | 3
  At least one serious AE | 0 | 0 | 0 | 0
  Discontinued study medication due to AE | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Whose Standard Deviation of Lateral Position (SDLP) Following Active Treatment As Compared to Placebo In Relation To The 2.5 cm SDLP Threshold
Description: SDLP was measured by an infrared camera mounted on the car's roof during a highway driving test. Lateral position of the car relative to the left lane boundary was recorded. The data summarizes the number of participants whose driving performance was worse, neutral or improved as compared to placebo at the 2.5 cm threshold. A neutral driving performance shows a difference of SDLP >= 2.5 cm and <= -2.5 cm when compared to placebo. A worse performance is when the difference of SDLP > 2.5 cm, and an improved performance is when the difference of SDLP < -2.5 cm.
Time Frame: 3-9 hours post dose
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Zolpidem 4 Hours Prior | Zolpidem 3 Hours Prior | Zopiclone
Number analyzed (Participants) | 40 | 40 | 40
participants
  Impaired | 5 | 10 | 18
  Neutral | 34 | 29 | 22
  Improved | 1 | 1 | 0

5. Primary Outcome: Probability of Differences From Placebo Exceeding The 2.5 cm Threshold in Standard Deviation of Lateral Position (SDLP) Following Administration of Active Therapy
Description: This table represents the probability of driving performance changes summarized in the previous table. It answers the question: What is the chance that # participants out of the total number of participants had better (or worse) driving performance? Probability values of <.001 are listed in the data table as 0.000.
  A symmetry analysis was conducted for the probability of difference in mean SDLP (treatment) - mean SDLP (placebo) exceeding thresholds. Statistically significant asymmetries indicate a decrement in driving performance.
Time Frame: 3-9 hours post dose
Population: Intent to treat population
Measure: Number; unit: proportion
Arm/Group | Zolpidem 4 Hours Prior | Zolpidem 3 Hours Prior | Zopiclone | Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40
proportion
  Probability - impaired | 0.125 | 0.250 | 0.450 | NA — Probability for the active treatment arms uses the Placebo experience as a base case from which to calculate probability.
  Probability - improved | 0.025 | 0.025 | 0.000 | NA — Probability for the active treatment arms uses the Placebo experience as a base case from which to calculate probability.
Statistical Analysis 1: Comparison: Zolpidem 4 Hours Prior vs Placebo; Symmetry analysis was performed for the probability of difference from placebo falling above and below the threshold of +/-2.5 cm in Standard Deviation of Lateral Position (SDLP) following administration of zolpidem tartrate sublingual tablet 4 hours prior to driving. Statistically significant asymmetries indicate a decrement in driving performance. Lack of statistical significance indicates symmetry which shows a lack of treatment effect on driving performance; Test type: Superiority or Other; p = 0.2188, McNemar — No adjustments. The a priori threshold for statistical significance is 0.05; McNemar's exact test with one degree of freedom is used
Statistical Analysis 2: Comparison: Zolpidem 3 Hours Prior vs Placebo; Symmetry analysis was performed for the probability of difference from placebo falling above and below the threshold of +/-2.5 cm in Standard Deviation of Lateral Position (SDLP) following administration of zolpidem tartrate sublingual tablet 3 hours prior to driving. Statistically significant asymmetries indicate a decrement in driving performance. Lack of statistical significance indicates symmetry which shows a lack of treatment effect on driving performance; Test type: Superiority or Other; p = 0.0117, McNemar — No adjustments. The a priori threshold for statistical significance is 0.05; McNemar's exact test with one degree of freedom is used
Statistical Analysis 3: Comparison: Zopiclone vs Placebo; Symmetry analysis was performed for the probability of difference from placebo falling above and below the threshold of +/-2.5 cm in Standard Deviation of Lateral Position (SDLP) following administration of zopiclone 9 hours prior to driving. Statistically significant asymmetries indicate a decrement in driving performance. Lack of statistical significance indicates symmetry which shows a lack of treatment effect on driving performance; Test type: Superiority or Other; p < 0.0001, McNemar — No adjustments. The a priori threshold for statistical significance is 0.05; McNemar's exact test with one degree of freedom is used

6. Secondary Outcome: Number of Participants Whose Standard Deviation of Lateral Position (SDLP) Following Active Treatment As Compared to Placebo In Relation To The 2.0 cm SDLP Threshold
Description: SDLP was measured by an infrared camera mounted on the car's roof during a highway driving test. Lateral position of the car relative to the left lane boundary was recorded. The data summarizes the number of participants whose driving performance was worse, neutral or improved as compared to placebo at the 2.0 cm threshold. A neutral driving performance shows a difference of SDLP >= 2.0 cm and <= -2.0 cm when compared to placebo. A worse performance is when the difference of SDLP > 2.0 cm, and an improved performance is when the difference of SDLP < -2.0 cm.
Time Frame: 3-9 hours post dose
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Zolpidem 4 Hours Prior | Zolpidem 3 Hours Prior | Zopiclone
Number analyzed (Participants) | 40 | 40 | 40
participants
  Impaired | 6 | 13 | 19
  Neutral | 33 | 25 | 21
  Improved | 1 | 2 | 0

7. Secondary Outcome: Probability of Differences From Placebo Exceeding The 2.0 cm Threshold in Standard Deviation of Lateral Position (SDLP) Following Administration of Active Therapy
Description: as for outcome 5
Time Frame: 3-9 hours post dose
Population: Intent to treat population
Measure: Number; unit: proportion
Arm/Group | Zolpidem 4 Hours Prior | Zolpidem 3 Hours Prior | Zopiclone | Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40
proportion
  Probability - impaired | 0.150 | 0.325 | 0.475 | NA — Probability for the active treatment arms uses the Placebo experience as a base case from which to calculate probability.
  Probability - improved | 0.025 | 0.050 | 0.000 | NA — Probability for the active treatment arms uses the Placebo experience as a base case from which to calculate probability.
Statistical Analysis 1: Comparison: Zolpidem 4 Hours Prior vs Placebo; Symmetry analysis was performed for the probability of difference from placebo falling above and below the threshold of +/-2.0 cm in Standard Deviation of Lateral Position (SDLP) following administration of zolpidem tartrate sublingual tablet 4 hours prior to driving. Statistically significant asymmetries indicate a decrement in driving performance. Lack of statistical significance indicates symmetry which shows a lack of treatment effect on driving performance; Test type: Superiority or Other; p = 0.1250, McNemar — No adjustments. The a priori threshold for statistical significance is 0.05; McNemar's exact test with one degree of freedom is used
Statistical Analysis 2: Comparison: Zolpidem 3 Hours Prior vs Placebo; Symmetry analysis was performed for the probability of difference from placebo falling above and below the threshold of +/-2.0 cm in Standard Deviation of Lateral Position (SDLP) following administration of zolpidem tartrate sublingual tablet 3 hours prior to driving. Statistically significant asymmetries indicate a decrement in driving performance. Lack of statistical significance indicates symmetry which shows a lack of treatment effect on driving performance; Test type: Superiority or Other; p = 0.0074, McNemar — No adjustments. The a priori threshold for statistical significance is 0.05; McNemar's exact test with one degree of freedom is used
Statistical Analysis 3: Comparison: Zopiclone vs Placebo; Symmetry analysis was performed for the probability of difference from placebo falling above and below the threshold of +/-2.0 cm in Standard Deviation of Lateral Position (SDLP) following administration of Zopiclone 9 hours prior to driving. Statistically significant asymmetries indicate a decrement in driving performance. Lack of statistical significance indicates symmetry which shows a lack of treatment effect on driving performance; Test type: Superiority or Other; p < 0.0001, McNemar — No adjustments. The a priori threshold for statistical significance is 0.05; McNemar's exact test with one degree of freedom is used

8. Secondary Outcome: Number of Participants Whose Standard Deviation of Lateral Position (SDLP) Following Active Treatment As Compared to Placebo In Relation To The 3.5 cm SDLP Threshold
Description: SDLP was measured by an infrared camera mounted on the car's roof during a highway driving test. Lateral position of the car relative to the left lane boundary was recorded. The data summarizes the number of participants whose driving performance was worse, neutral or improved as compared to placebo at the 3.5 cm threshold. A neutral driving performance shows a difference of SDLP >= 3.5 cm and <= -3.5 cm when compared to placebo. A worse performance is when the difference of SDLP > 3.5 cm, and an improved performance is when the difference of SDLP < -3.5 cm.
Time Frame: 3-9 hours post dose
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Zolpidem 4 Hours Prior | Zolpidem 3 Hours Prior | Zopiclone
Number analyzed (Participants) | 40 | 40 | 40
participants
  Impaired | 2 | 7 | 14
  Neutral | 38 | 33 | 26
  Improved | 0 | 0 | 0

9. Secondary Outcome: Probability of Differences From Placebo Exceeding The 3.5 cm Threshold in Standard Deviation of Lateral Position (SDLP) Following Administration of Active Therapy
Description: as for outcome 5
Time Frame: 3-9 hours post dose
Population: Intent to treat population
Measure: Number; unit: proportion
Arm/Group | Zolpidem 4 Hours Prior | Zolpidem 3 Hours Prior | Zopiclone | Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40
proportion
  Probability - impaired | 0.050 | 0.175 | 0.350 | NA — Probability for the active treatment arms uses the Placebo experience as a base case from which to calculate probability.
  Probability - improved | 0.000 | 0.000 | 0.000 | NA — Probability for the active treatment arms uses the Placebo experience as a base case from which to calculate probability.
Statistical Analysis 1: Comparison: Zolpidem 4 Hours Prior vs Placebo; Symmetry analysis was performed for the probability of difference from placebo falling above and below the threshold of +/-3.5 cm in Standard Deviation of Lateral Position (SDLP) following administration of zolpidem tartrate sublingual tablet 4 hours prior to driving. Statistically significant asymmetries indicate a decrement in driving performance. Lack of statistical significance indicates symmetry which shows a lack of treatment effect on driving performance; Test type: Superiority or Other; p = 0.5000, McNemar — No adjustments. The a priori threshold for statistical significance is 0.05; McNemar's exact test with one degree of freedom is used
Statistical Analysis 2: Comparison: Zolpidem 3 Hours Prior vs Placebo; Symmetry analysis was performed for the probability of difference from placebo falling above and below the threshold of +/-3.5 cm in Standard Deviation of Lateral Position (SDLP) following administration of zolpidem tartrate sublingual tablet 3 hours prior to driving. Statistically significant asymmetries indicate a decrement in driving performance. Lack of statistical significance indicates symmetry which shows a lack of treatment effect on driving performance; Test type: Superiority or Other; p = 0.0156, McNemar — No adjustments. The a priori threshold for statistical significance is 0.05; McNemar's exact test with one degree of freedom is used
Statistical Analysis 3: Comparison: Zopiclone vs Placebo; Symmetry analysis was performed for the probability of difference from placebo falling above and below the threshold of +/-3.5 cm in Standard Deviation of Lateral Position (SDLP) following administration of zopiclone 9 hours prior to driving. Statistically significant asymmetries indicate a decrement in driving performance. Lack of statistical significance indicates symmetry which shows a lack of treatment effect on driving performance; Test type: Superiority or Other; p = 0.0001, McNemar — No adjustments. The a priori threshold for statistical significance is 0.05; McNemar's exact test with one degree of freedom is used

ADVERSE EVENTS:
Time Frame: Treatment emergent AEs (Day 1 to Week 6)
Arm/Group | Zolpidem 4 Hours Prior | Zolpidem 3 Hours Prior | Zopiclone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 5/40 | 5/40 | 6/40 | 4/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolpidem 4 Hours Prior (N=40) | Zolpidem 3 Hours Prior (N=40) | Zopiclone (N=40) | Placebo (N=40)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
No studies directly connect SDLP thresholds with an increased risk of an accident for an individual. Nor has a SDLP threshold been adopted by a regulatory body. Based on published literature, an SDLP change of 2.5 cm was used in the primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor agrees to review manuscripts within a reasonable period of time. If sponsor determines the publication included patentable subject matter, sponsor will be granted no less than 120 days to prepare patent applications.